CLINICAL TRIAL: NCT03890809
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of BMS-986165 in Participants With Normal Hepatic Function and Participants With Mild, Moderate and Severe Hepatic Impairment
Brief Title: An Investigational Study of BMS-986165 in Participants With Normal Liver Function and Participants With Mild to Severe Liver Damage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-062; 2018-002534-20 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Liver Dysfunction; Healthy Volunteers
MeSH Terms: conditions — Liver Diseases | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Normal liver function (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Mild liver impairment (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Moderate liver impairment (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Severe liver impairment (Experimental): Single dose
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral administration

SUMMARY:
The purpose of this study is to investigate BMS-986165 in participants with different levels of liver function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body mass index of 18.0 to 38.0 kg/m2, inclusive, and weight ≥ 50 kg, at screening
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) > 80 mL/min/1.73 m2 for participants

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the participant
* History or clinical evidence of acute or chronic bacterial infection (eg, pneumonia, septicemia) within 3 months prior to screening
* Have a history of cancer (malignancy) with the following exceptions: (1) participants with adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the trial; (2) participants with other malignancies who have been successfully treated ≥10 years prior to the screening visit where, in the judgment of both the investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the screening visit

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Approximately 9 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | Approximately 9 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Approximately 9 days

SECONDARY OUTCOMES:
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | Approximately 44 days
Number of clinically significant changes in clinical laboratory values, vital signs, ECGs, and physical examinations | Approximately 44 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Pharmaceutical Research Associates CZ, s.r.o, Prague, Czechia
- Hungary (2):
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
  - Clinical Research Unit Hungary, Miskolc
- Local Institution, Bratislava, Slovakia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm